CLINICAL TRIAL: NCT05153330
Title: A Phase 1 First-in-human Dose-escalation and Dose-expansion Study of BMF-219, an Oral Covalent Menin Inhibitor, in Adult Patients With Acute Leukemia (AL), Diffuse Large B-cell Lymphoma (DLBCL), Multiple Myeloma (MM), and Chronic Lymphocytic Leukemia (CLL)/ Small Lymphocytic Lymphoma (SLL)
Brief Title: Study of BMF-219, a Covalent Menin Inhibitor, in Adult Patients With AML, ALL (With KMT2A/ MLL1r, NPM1 Mutations), DLBCL, MM, and CLL/SLL
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Biomea Fusion, Inc., is no longer pursuing oncology indications for BMF-219. No safety concerns or efficacy observations led to this study closure.
Sponsor: Biomea Fusion Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVALENT-101
Record Dates: First submitted 2021-11-30; First posted 2021-12-10 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Acute Mixed-Phenotype Leukemia; Cancer; Refractory; Progression; Diffuse Large B Cell Lymphoma; Multiple Myeloma; Lymphoma; Lymphoma, Non-Hodgkin; Myeloma, Plasma-Cell; Myelomatosis; Plasma Cell Myeloma; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasms; Disease Progression; Lymphoma, Large B-Cell, Diffuse; Multiple Myeloma; Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Intervention Model Description: The first-in-human (FIH) study is a dose-escalation/dose-expansion study of BMF-219. During the dose-escalation phase of the study, the optimal biologic dose (OBD) and recommended Phase 2 dose (RP2D) of BMF-219 will be determined. Subjects in Cohort 1 (acute leukemia) are assigned to one of two parallel arms; ARM A (subjects not receiving CYP3A4 inhibitors) and ARM B (subjects receiving CYP3A4 inhibitors); Subjects in Cohort 2 (DLBCL), Cohort 3 (multiple myeloma), and Cohort 4 (chronic lymphocytic leukemia/ small lymphocytic lymphoma) are assigned to a single arm (ARM A).The dose-expansion phase will obtain further safety, as well as efficacy data for BMF-219 when dosed at the OBD and RP2D.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Experimental): Experimental: ARM A:
  Study participants who are not receiving a moderate or strong CYP3A4 inhibitor.
  Dose Escalation Phase:
  * Cohort 1: Participants with acute leukemia
  * Cohort 2: Participants with diffuse large B-cell lymphoma
  * Cohort 3: Participants with multiple myeloma
  * Cohort 4: Participants with chronic lymphocytic leukemia/ small lymphocytic lymphoma
  Participants will receive escalating dose BMF-219 orally once per day to identify the OBD/RP2D (Optimal Biologic Dose/Recommended Ph2 Dose).
  Dose Expansion Phase:
  Cohorts 1, 2, 3, and 4 will receive BMF-219 at the OBD/ RP2D to further assess the safety/ efficacy of the investigational drug.
  Interventions: Drug: BMF-219
- Dose Expansion (Experimental): Experimental: ARM B:
  Study participants who are receiving a moderate or strong CYP3A4 inhibitor.
  Dose Escalation Phase:
  • Cohort 1: Participants with acute leukemia will receive escalating dose BMF-219 orally to identify the OBD/ RP2D (Optimal Biologic Dose/Recommended Ph2 Dose).
  Dose Expansion Phase:
  Cohort 1 will receive BMF-219 at the OBD/ RP2D to further assess the safety and efficacy of the investigational drug.
  Interventions: Drug: BMF-219

INTERVENTIONS:
Drug: BMF-219 — BMF-219 is orally administered in continuous 28 day cycles. Alternative BID dosage may be used.
  Other Names: Covalent Menin Inhibitor

SUMMARY:
A Phase 1 first-in-human dose-escalation and dose-expansion study of BMF-219, an oral covalent menin inhibitor, in adult patients with AML, ALL (with KMT2A/ MLL1r, NPM1 mutations), DLBCL, MM, and CLL/SLL.

DETAILED DESCRIPTION:
A Phase 1 first-in-human dose-escalation and dose-expansion study of BMF-219, an oral covalent menin inhibitor, in adult patients with acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL) with mixed lineage leukemia 1-rearranged (KMT2A/ MLL1r), nucleophosmin 1 (NPM1), diffuse large b-cell lymphoma (DLBCL), multiple myeloma (MM), and chronic lymphocytic lymphoma (CLL)/ small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* All subjects must have histologically or pathologically confirmed diagnosis of their malignancy and/ or measurable R/ R disease, as follows:

  1. Cohort 1 only: Refractory or relapsed acute leukemia defined as > 5% blasts in the bone marrow or reappearance of blasts in the peripheral blood.
  2. Cohort 2 only: Previously treated, pathologically confirmed de novo DLBCL, or DLBCL transformed from previously indolent lymphoma (e.g., follicular lymphoma) with documented clinical or radiological evidence of progressive or persistent disease. At study entry, subjects must have measurable disease as per the revised criteria for response assessment of lymphoma.
  3. Cohort 3 only: Measurable MM.
  4. Cohort 4 only: Previously treated subjects with active CLL/SLL with meeting at least 1 of the iwCLL 2018 criteria for requiring treatment.
* Subjects must be refractory or must have progressed on, or following discontinuation of the most recent anti-cancer therapy, with the following considerations:

  1. Cohort 1 only: Have failed or are ineligible for any approved standard of care therapies, including HSCT (Hematopoietic Stem Cell Transplantation).
  2. Cohort 2 only: Must have received at least 2 previous systemic regimens for the treatment of their de novo or transformed DLBCL.
  3. Cohort 3 only: Must have received at least 3 anti-MM regimens including proteasome inhibitor.
  4. Cohort 4 only: Must have received at least 2 prior systemic treatment regimens.
* ECOG performance status of 0-2 and an estimated expected life expectancy of > 3 months in the opinion of the Investigator.
* Adequate organ function.
* Both men and women of childbearing potential or their partners must use adequate birth control measures during the course of the trial and for at least 90 days after discontinuing study treatment.

Exclusion Criteria:

Subjects who meet any of the following criteria will not be enrolled in the study (all cohorts, unless otherwise indicated):

* Certain disease subtypes or occurrences, as follows:

  1. Cohort 1: Acute promyelocytic leukemia (APL), chronic myeloid leukemia (CML) in blast crisis.
  2. Cohort 2: Primary mediastinal B-cell lymphoma (PMBCL), DLBCL transformed from diseases other than indolent non-Hodgkin's Lymphoma (NHL).
  3. Cohort 3: Active plasma cell leukemia, myeloma with amyloidosis, systemic light chain amyloidosis.
  4. Cohort 4: Known or suspected history of Richter's transformation.
* White Blood Count (WBC) > 50,000/μL (uncontrollable with cytoreductive therapy) (Cohort 1 only).
* Known central nervous involvement, as follows:

  1. Cohort 1: Clinically active central nervous system (CNS) leukemia. Previously controlled CNS leukemia is acceptable.
  2. Cohort 2: Active CNS lymphoma or meningeal involvement.
  3. Cohort 3: Active CNS MM.
  4. Cohort 4: Active CNS leukemia.
* Prior menin inhibitor therapy.
* Known positive test for human immunodeficiency virus, hepatitis C, or hepatitis B surface antigen.
* Subjects with a pre-existing disorder predisposing them to a serious or life-threatening infection.
* An active uncontrolled acute or chronic systemic fungal, bacterial, or viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-05-02 (Actual)

PRIMARY OUTCOMES:
Determine Optimal Biologic Dose (OBD) and RP2D of BMF-219 monotherapy for (Cohorts 1, 2, 3 & 4) | At the end of Cycle 1 (each Cycle is 28 Days in duration)
  Determine Optimal Biologic Dose (OBD) and recommended Phase 2 dose (RP2D) of BMF-219 monotherapy in subjects with refractory or relapsed (R/ R) acute leukemia (Cohort 1), diffuse large B-cell lymphoma (Cohort 2), multiple myeloma (Cohort 3), and chronic lymphocytic leukemia/ small lymphocytic lymphoma (Cohort 4).

SECONDARY OUTCOMES:
Evaluate the Safety treatment-emergent TEAEs and SAEs | 28 Days after last dose.
  Evaluate the Safety of BMF-219 as expressed by treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Steve Morris, MD, Study Director — Biomea Fusion Inc.
Locations (41):
- United States (17):
  - University of California, Irvine, Irvine, California
  - University of Southern California Norris Cancer Center, Los Angeles, California
  - UCLA Department of Medicine, Los Angeles, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Stanford Cancer Center, Stanford, California
  - Mayo Clinic, Jacksonville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Blood & Marrow Transplant Group of GA (Northside Hospital), Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Henry Ford Hospital, Detroit, Michigan
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Gainesville, Virginia
- Greece (2):
  - Evangelismos General Hospital of Athens, Athens
  - Alexandra General Hospital of Athens, Athens
- Italy (7):
  - AOU Ospedali Riuniti Ancona, Ancona
  - ASST Papa Giovanni XXIII Hospital Bergamo, Bergamo
  - Instituto Clinico Humanitas, Milan
  - IRCCS Ospedale San Raffaele, Programma di Ricerca Strategica su LLC, Milan
  - Istituto Europeo di Oncologia, Milan
  - Ospedale Santa Maria della Misericordia, Perugia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Netherlands (4):
  - Amsterdam UMC, Amsterdam
  - UMCG Groningen, Groningen
  - Radboud University Medical Center, Nijmegen
  - Erasmus University Medical Center Rotterdam, Rotterdam
- Spain (11):
  - Hospital General de Albacete, Albacete
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No